CLINICAL TRIAL: NCT07386561
Title: Adjunctive Virtual Reality Therapy Versus Non-Sleep Deep Rest Relaxation During Postoperative Rehabilitation in Older Adults Undergoing Hip or Knee Arthroplasty
Brief Title: Virtual Reality Therapy and Non-Sleep Deep Rest Relaxation After Joint Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Wroclaw Medical University (Other); Jan Dlugosz University in Czestochowa (Other)
Responsible Party: Principal Investigator, Joanna Szczepańska-Gieracha, Principal Investigator, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KE-U/108/2025
Record Dates: First submitted 2026-01-26; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Arthropathy; Osteoarthritis, Hip; Osteoarthritis, Knee
Keywords: virtual reality; arthroplasty; psychological outcomes; functional state; anxiety; stress; ortopedic rehabilitation; relaxation
MeSH Terms: conditions — Joint Diseases; Osteoarthritis, Hip; Osteoarthritis, Knee; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immersive Virtual Reality Therapy Group (Experimental): Conventional orthopedic rehabilitation supplemented by VR therapy
  Interventions: Device: Immersive Virtual Reality Therapy; Behavioral: Conventional rehabilitation
- NSDR Group (Experimental): Conventional orthopedic rehabilitation supplemented by non-sleep deep rest relaxation
  Interventions: Behavioral: Non-Sleep Deep Rest Relaxation; Behavioral: Conventional rehabilitation
- Conventional Rehabilitation Group (Active Comparator): Conventional orthopedic rehabilitation
  Interventions: Behavioral: Conventional rehabilitation

INTERVENTIONS:
Device: Immersive Virtual Reality Therapy — 8 sessions of VR therapy over 4 weeks (each of them 20 minutes long). As a virtual reality source, VRTierOne device (Stolgraf®) were used. Thanks to using head mounted display and the phenomenon of total immersion VR therapy provides an intense visual, auditory and kinesthetic stimulation. It can have a calming and mood-improving effect or help the patients recognize their psychological resources and motivate to the rehabilitation process. In the virtual therapeutic garden there are a rich set of symbols and metaphors based on Ericksonian Psychotherapy approach. The most important is the Garden of Revival which symbolizes the patient's health. It used to be full of life and energy, now it is neglected, requires work to be revived. In the therapeutic process day by day, the therapist tells the patient a symbolic story about his/her situation.
  Arms: Immersive Virtual Reality Therapy Group
Behavioral: Non-Sleep Deep Rest Relaxation — The experimental group will receive eight sessions of audio recording based on the Non-Sleep Deep Rest (NSDR) concept during the 4-week rehabilitation program. Each 20-minute session is conducted in a quiet setting using noisecancelling headphones. The recording guides patients through a structured body scan, directing attention sequentially to specific body regions and prompting active muscle relaxation. Body scanning is combined with mindful breathing to deepen relaxation and attenuate sympathetic nervous system activity. Therapeutic suggestions focus on reframing overload versus relief, letting go versus holding on, and balancing action with awareness. The intervention aims to enhance psychological resilience and support the balance between the sympathetic and parasympathetic parts of the autonomic nervous system. The protocol is non-invasive, safe, and feasible for routine clinical use.
  Arms: NSDR Group
Behavioral: Conventional rehabilitation — Conventional rehabilitation follows standard postoperative protocols after hip or knee arthroplasty. The 4-week program includes five weekly sessions. Gait training is conducted in hospital corridors under physiotherapist supervision, using assistive devices as needed (crutches, walkers). Daily therapy includes 120 minutes of kinesiotherapy (general exercises and gait training), 30 minutes of ergotherapy to improve functional independence, and three individualized physical therapy procedures (laser therapy, magnetic therapy, or electrotherapy) tailored to patient needs.

SUMMARY:
The aim of this study is to compare the effectiveness of Virtual Reality therapy (VR therapy), Non-Sleep Deep Rest relaxation (NSDR relaxation) each delivered as an adjunct to standard postoperative rehabilitation, in older adults following hip or knee arthroplasty, focusing on reducing psychological stress and improving functional recovery.

DETAILED DESCRIPTION:
Older adults undergoing hip or knee arthroplasty frequently experience psychological distress, including elevated stress and anxiety, which may reduce engagement in rehabilitation and limit functional recovery. This randomized clinical trial will compare the effectiveness of Virtual Reality therapy (VR therapy) and Non-Sleep Deep Rest relaxation (NSDR relaxation) each delivered as an adjunct to standard postoperative rehabilitation, in this population. Ninety participants aged 60-85 years, within three months post-arthroplasty, will be recruited from an inpatient rehabilitation unit and randomized to receive standard rehabilitation alone, standard rehabilitation plus VR therapy or standard rehabilitation plus NSDR relaxation over a four-week period. The VR therapy will consist of eight 20-minute session using VRTierOne medical device. NSDR relaxation will be delivered as eight 20-minute, audio-guided relaxation sessions (body scan and breathing exercises) via noise-cancelling headphones in a quiet environment. Primary outcomes will include changes in psychological distress (stress, anxiety, depressive symptoms; assessed with validated questionnaires) and functional recovery (functional performance and mobility indices), measured at baseline and post-intervention. Both adjuncts are designed to be safe, well-tolerated, and feasible for clinical implementation. The findings are expected to clarify the comparative role of VR therapy and NSDR relaxation as low-risk adjunctive strategies to support psychological well-being and functional outcomes during post-arthroplasty rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 60 years and above who have recently (within the past 3 months) undergone knee or hip joint arthroplasty surgery.

Exclusion Criteria:

* Hearing impairment preventing the use of audio recordings;
* Cognitive impairment precluding independent completion of study questionnaires;
* History of disorders of consciousness, psychotic symptoms, bipolar disorder, or other severe psychiatric disorders;
* Current use of psychoactive medications;
* Ongoing psychiatric treatment or participation in individual psychological therapy;
* Functional status precluding independent ambulation (e.g., wheelchair-bound or bedridden; use of orthopedic aids such as crutches or a walker is permitted);
* Withdrawal of consent or refusal to participate at any stage of the study.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hospital Anxiety and Depression Scale (HADS) Score at 4 Weeks | Baseline and 4 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item instrument assessing anxiety and depression symptoms in hospital patients. Each item is scored from 0 to 3, with total scores ranging from 0 to 42. Higher scores indicate greater symptom severity.
Change from Baseline in Perceived Stress Scale (PSS-10) Score at 4 Weeks | Baseline and 4 weeks
  The Perceived Stress Scale (PSS-10) is a 10-item scale measuring perceived stress over the past month. Scores range from 0 to 40, with higher scores reflecting greater perceived stress.
Change from Baseline in Generalized Self-Efficacy Scale (GSES) Score at 4 Weeks | Baseline and 4 weeks
  The Generalized Self-Efficacy Scale (GSES) is a 10-item measure of general self-efficacy, meaning a person's broad belief in their ability to cope with difficult demands and handle challenges. Items are rated on a 4-point scale and summed to a total score ranging from 10 to 40. Higher scores reflect greater generalized self-efficacy.
Change from Baseline in Perception of Stress Questionnaire (PSQ) Score at 4 Weeks | Baseline and 4 weeks
  The Perception of Stress Questionnaire (PSQ) is a 27-item measure of perceived stress, with scores ranging from 21 to 105. Higher scores reflect greater stress perception.

SECONDARY OUTCOMES:
Change from Baseline in Rivermead Mobility Index (RMI) Score at 4 Weeks | Baseline and 4 weeks
  The Rivermead Mobility Index (RMI) consists of 14 items evaluating mobility tasks, with scores ranging from 0 (unable) to 14 (full mobility). Higher scores indicate better mobility.
Change from Baseline in Short Physical Performance Battery (SPPB) Score at 4 Weeks | Baseline and 4 weeks
  The Short Physical Performance Battery (SPPB) combines assessments of balance, gait speed, and chair stand tests, with composite scores ranging from 0 (worst) to 12 (best). Higher scores indicate better physical function.
Change from Baseline in Barthel Index Score at 4 Weeks | Baseline and 4 weeks
  The Barthel Index assesses independence in activities of daily living (ADL), with scores ranging from 0 to 100. Higher scores represent greater functional independence.
Change from Baseline in Tinetti's Short Scale Score at 4 Weeks | Baseline and 4 weeks
  Tinetti's Short Scale assesses fall risk through evaluation of gait and balance over five tasks. Scores range from 0 to 15, with higher scores indicating better functional mobility.
Change from Baseline in Visual Analogue Scale (VAS) Score at 4 Weeks | Baseline and 4 weeks
  The Visual Analogue Scale (VAS) is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured, commonly used to assess pain intensity. The scale consists of a 10 cm (100 mm) horizontal line, with endpoints defining extreme limits such as "no pain" and "worst pain imaginable." The patient marks a point on the line that represents their current state. Scores range from 0 to 100 mm, with higher scores indicating greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Szczepańska-Gierahca, PhD, Principal Investigator — Wrocław University of Health and Sport Sciences; Justyna Mazurek, PhD, Principal Investigator — Wroclaw Medical University; Błażej Cieślik, PhD, Principal Investigator — Jan Dlugosz University in Czestochowa
Locations (1):
- St. Hedwig of Silesia Hospital in Trzebnica, Trzebnica, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No